CLINICAL TRIAL: NCT00857428
Title: A Study to Evaluate the Relative Bioavailability of Oxymorphone 40 mg Extended-Release Tablets (Sandoz, Inc.) Compared to Opana ER (Oxymorphone Hydrochloride) Extended-Release Tablets, 40 mg (Endo Pharmaceuticals, Inc.) in Healthy Volunteers Under Fasted Conditions
Brief Title: Bioavailability of Oxymorphone Hydrochloride 40 mg Extended Release Tablets Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP Product Development, Sandoz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10713409
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oxymorphone ER 40 mg tablets Sandoz
  Interventions: Drug: oxymorphone
- 2 (Active Comparator): Opana ER 40 mg tablets Eon Pharmaceuticals
  Interventions: Drug: Oxymorphone

INTERVENTIONS:
Drug: oxymorphone — Tablets
  Other Names: Opana
  Arms: 1
Drug: Oxymorphone — 40 mg tablets
  Other Names: Opana
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioequivalence of oxymorphone hydrochloride extended-release tablets (Sandoz) with Opana extended release oxymorphone hydrochloride tablets.

DETAILED DESCRIPTION:
Bioequivalence based on FDA Criteria.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, medical history or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C
* Treatment for drug or alcohol dependence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC | Four Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daryl G. Ficklin, D.O., Principal Investigator — Novum Pharmaceutical Research Services